CLINICAL TRIAL: NCT03035162
Title: Dual-hemisphere Transcranial Direct Current Stimulation on Lower Limb Motor Functions After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Wanalee Klomjai, Principal Investigator, Mahidol University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MU-CIRB 2016/048.0704
Record Dates: First submitted 2017-01-25; First posted 2017-01-27 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Stroke
Keywords: dual tDCS; physical rehabilitation; lower limb functions
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS & PT (Experimental): Dual transcranial direct current stimulation (tDCS) will be applied over the leg motor area (M1) priori to conventional physical therapy (1 hours). Anodal on affected hemisphere, Cathodal on unaffected hemisphere. Current intensity is fixed at 2 mA and current will flow continuously during 20 minutes for the active conditions. Physical therapist will give an intervention program exactly the same in all cases. The scope of intervention is administered to improve strength of weakened and postural lower limbs muscles such as trunk muscles, hip flexors/extensors/abductors, knee flexors/extensors.
  Interventions: Device: Transcranial direct current stimulation
- Sham tDCS & PT (Active Comparator): Dual transcranial direct current stimulation (tDCS) will be applied over the leg motor area (M1) priori to conventional physical therapy (1 hours). Anodal on affected hemisphere, Cathodal on unaffected hemisphere. Current intensity is fixed at 2 mA and current will flow only 2 minutes for the sham conditions. Physical therapist will give an intervention program exactly the same in all cases. The scope of intervention is administered to improve strength of weakened and postural lower limbs muscles such as trunk muscles, hip flexors/extensors/abductors, knee flexors/extensors.
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — Dual Active/sham tDCS will be applied over the leg motor area (M1) priori to conventional physical therapy (1 hours). Anodal on affected hemisphere, Cathodal on unaffected hemisphere. Each participant will complete two experiments (active/sham tDCS). The interval between two experiments is at least 48 hours. The two experiments will be performed in random order for each subject.

SUMMARY:
The aim of the present study is to evaluate the possible effect of using dual-tDCS combined with conventional physical therapy on lower limb function in stroke patients.

DETAILED DESCRIPTION:
Stroke is a leading cause of adult motor disability. The recovery of motor function after stroke is often incomplete, despite classical rehabilitation techniques. In the beginning of the 21th century, transcranial direct current stimulation (tDCS) was introduced as a non-invasive tool to reversibly modulate brain excitability in humans in which a device sends constant low direct current (DC) delivered to the area of interest through the electrodes. These findings have opened the way to the therapeutic use of the brain stimulation for stroke. Based on the polarity-specific effects, anodal tDCS increases cortical excitability and cathodal tDCS decreases cortical excitability. To change the cortical excitability, tDCS differs from other brain stimulation techniques such as transcranial magnetic stimulation (TMS) in that it does not cause action potentials in cortical neurons, but rather induces shifts in neuronal resting membrane potential . This is considered to induce a lesser or no risk of a seizure. Given its advantages such as non-invasiveness, painlessness, safety, and possible after-effects, tDCS rapidly become a therapeutic adjuvant in neurorehabilitation especially in stroke patients with motor deficits . A number of studies in healthy subjects and stroke patients have reported that tDCS-induced excitability changes are related to increase in the performance of motor tasks and motor skills learning, mainly upper limb functions Recenty, dual-hemisphere tDCS in which, excites one hemisphere using anodal stimulation and inhibits the other by cathodal stimulation has been described in healthy subjects to greater enhance hand motor learning compared to uni-hemisphere tDCS. The corresponding tDCS-induced changes were reported in imaging study to involve interhemispheric interactions . An increase in the excitability of unaffected hemisphere and an abnormally high interhemispheric inhibition (IHI) drive from intact to lesioned hemisphere have been widely reported after unilateral stroke. Dual-tDCS has been more recent used in rehabilitation aiming to reduce the inhibition exerted by the unaffected hemisphere on the affected hemisphere and restore the normal balance of the IHI. Dual-tDCS combined with training or simultaneous occupational/physical therapy has been reported to improve motor skill learning and functions of the paretic upper limb in chronic stroke patients .

Lower-limb functions are commonly disordered after stoke, however, less study has focused the effect of tDCS on lower limb functions. A single session of anodal tDCS over the lower limb M1 has reported to acutely enhance the effect of motor practice of the paretic ankle, force production of the paretic knee extensors, and postural stability in chronic stroke patients. However, little is known about effects of dual-tDCS on lower limb in stroke patients. Only one recent study showed an improvement of walking speed immediately after a single session of dual-tDCS alone in sub-acute stroke patients .

ELIGIBILITY:
Inclusion Criteria:

1. Age range 18-75 years.
2. First ever-ischemic lesion in the territory of middle cerebral artery or anterior cerebral artery. CT scan/MRI result is thus required.
3. Sub acute phase of stroke (less than 6 months)
4. Able to sit-to-stand and stand-to-sit independently
5. Able to walk without physical assistance at least 6 m
6. Free of any neurological antecedent, unstable medical conditions or condition that may increase the risk of stimulation such as epilepsy; although tDCS is believed to induce less or no risk of seizure and epileptic seizure have never been reported in tDCS study even in a study with active epilepsy (Fregni et al., 2006).

Exclusion Criteria:

1. Pre-stroke disability
2. Pregnant
3. Be unable to understand the instruction
4. No clear neurological antecedent history or psychiatric disorder
5. Excessive pain in any joint of the paretic limb (numerical pain rating score > 7)
6. Presence of intracranial metal implantation, cochlea implant, or cardiac pacemaker
7. Subjects are participating in the other protocol or receiving alternative treatment such as acupuncture

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Strength | 15 minutes
  Knee extensors strength is required to perform lower functions including sit-to-stand and gait. Knee extensor strength will measure using Biodex system, performing while the subjects comfortably seat in the position of knee flexed at 120° and ankle at 110° of plantar flexion on the attached footplate. Subjects will perform 3 isometric maximum voluntary contraction (MVC) of the knee extensor during a duration of 5 sec, separated by 2 min rest. The highest MVC in each session will be used as MVC level.
Five-Times-Sit-To-Stand test (FTSST) | 5 minutes
  Subject will sits with arms folded across chest or the paretic arm at the side or in a sling. Subjects will be instructed as the following "I want you to stand up and sit down 5 times as quickly as you can when I say 'Go'." Subjects must be fully standing between repetitions. Timing will begin at "GO" and ends when the patient's buttocks touch the seat after the fifth sit-to-stand.
Timed Up & Go test (TUG) | 5 minutes
  Subjects will sits on the chair and place their back against the chair. Timing will begin at "GO", the subjects will be asked to walk 3m, turn, walk back, and sit down. The stopwatch stops when the patient's buttocks touch the seat.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty ofPhysical Therapy, Mahidol University, Salaya, Nakonpathom, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cabral ME, Baltar A, Borba R, Galvao S, Santos L, Fregni F, Monte-Silva K. Transcranial direct current stimulation: before, during, or after motor training? Neuroreport. 2015 Aug 5;26(11):618-22. doi: 10.1097/WNR.0000000000000397. PMID 26049257
- [Background] Fregni F, Thome-Souza S, Nitsche MA, Freedman SD, Valente KD, Pascual-Leone A. A controlled clinical trial of cathodal DC polarization in patients with refractory epilepsy. Epilepsia. 2006 Feb;47(2):335-42. doi: 10.1111/j.1528-1167.2006.00426.x. PMID 16499758
- [Background] Jeffery DT, Norton JA, Roy FD, Gorassini MA. Effects of transcranial direct current stimulation on the excitability of the leg motor cortex. Exp Brain Res. 2007 Sep;182(2):281-7. doi: 10.1007/s00221-007-1093-y. Epub 2007 Aug 24. PMID 17717651
- [Background] Kim CR, Kim DY, Kim LS, Chun MH, Kim SJ, Park CH. Modulation of cortical activity after anodal transcranial direct current stimulation of the lower limb motor cortex: a functional MRI study. Brain Stimul. 2012 Oct;5(4):462-7. doi: 10.1016/j.brs.2011.08.002. Epub 2011 Aug 26. PMID 21962977
- [Background] Nitsche MA, Paulus W. Excitability changes induced in the human motor cortex by weak transcranial direct current stimulation. J Physiol. 2000 Sep 15;527 Pt 3(Pt 3):633-9. doi: 10.1111/j.1469-7793.2000.t01-1-00633.x. PMID 10990547
- [Background] Roche N, Lackmy A, Achache V, Bussel B, Katz R. Effects of anodal transcranial direct current stimulation over the leg motor area on lumbar spinal network excitability in healthy subjects. J Physiol. 2011 Jun 1;589(Pt 11):2813-26. doi: 10.1113/jphysiol.2011.205161. Epub 2011 Apr 18. PMID 21502292
- [Background] Roche N, Lackmy A, Achache V, Bussel B, Katz R. Effects of anodal tDCS on lumbar propriospinal system in healthy subjects. Clin Neurophysiol. 2012 May;123(5):1027-34. doi: 10.1016/j.clinph.2011.09.011. Epub 2011 Oct 20. PMID 22014699